CLINICAL TRIAL: NCT01440816
Title: A Phase II Study of Intratumoral Injection of Interleukin-12 Plasmid and in Vivo Electroporation in Patients With Merkel Cell Carcinoma
Brief Title: IL-12 Gene and in Vivo Electroporation-Mediated Plasmid DNA Vaccine Therapy in Patients With Merkel Cell Cancer
Acronym: MCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OncoSec Medical Incorporated (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMS-I110; NCI-2011-01221 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH)
Record Dates: First submitted 2011-09-23; First posted 2011-09-27 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A: Tavo-EP (Experimental): Patients in Cohort A received one cycle (3 daily treatments on Days 1, 5, and 8) of intra-tumoral injection(s) of tavo at a fixed dose of 0.5 mg/mL (up to 4 tumor sites) followed immediately by in vivo electroporation, after which they proceeded to definitive treatment (surgery and/or radiation therapy) which started between 2 and 4 weeks after the first injection.
  Interventions: Biological: Tavokinogene Telseplasmid (tavo); Device: OncoSec Medical System (OMS)
- Cohort B: Tavo-EP (Experimental): Patients in Cohort B received up to 4 cycles (3 daily treatments on Days 1, 5, and 8, per cycle) of intra-tumoral injection(s) of tavo at a fixed dose of 0.5 mg/mL (up to 4 tumor sites) followed immediately by in vivo electroporation, with 12 planned weeks between each cycle, lasting up to 12 months.
  Interventions: Biological: Tavokinogene Telseplasmid (tavo); Device: OncoSec Medical System (OMS)

INTERVENTIONS:
Biological: Tavokinogene Telseplasmid (tavo) — Patients received intratumoral injection(s) of tavo.
  Other Names: interleukin-12 gene; IL-12 gene; pIL-12; plasmid DNA encoding human interleukin-12; plasmid IL-12
Device: OncoSec Medical System (OMS) — Electroporation via OMS was performed immediately following intratumoral injection of tavo. A sterile applicator containing 6 stainless steel electrodes arranged in a circle were placed around the tumor. The applicator was connected to the OMS power supply and six pulses were administered to each tumor lesion at the approximate point of tavo injection.
  Other Names: MedPulser

SUMMARY:
This phase II trial studies the effectiveness of ImmunoPulse IL-12® in treating patients with Merkel cell cancer. ImmunoPulse IL-12® is the combination of intratumoral interleukin-12 gene (also known as tavokinogene telseplasmid [tavo]) and in vivo electroporation-mediated plasmid deoxyribonucleic acid [DNA] vaccine therapy (tavo-EP) administered using the OncoSec Medical System (OMS). Placing the gene for interleukin-12 into Merkel cells may help the mount an effective anti-tumor immune response to kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To measure the effect of intratumoral injection of tavo followed by in vivo electroporation (EP) (electroporation-mediated plasmid DNA vaccine therapy) on the local expression of interleukin-12 (IL-12) in the tumor microenvironment in patients with Merkel cell carcinoma (MCC).

SECONDARY OBJECTIVES:

I. To assess the safety of tavo-EP in MCC. II. To assess the clinical efficacy of this treatment approach in MCC. III. To assess the immunologic changes resulting from this treatment approach.

OUTLINE:

Patients receive tavo intratumorally (IT) and undergo electrical discharge via OMS around the tumor site for electroporation-mediated plasmid DNA vaccine therapy on days 1, 5, and 8. Patients with unresectable disease may receive a second course of treatment in 12 weeks. Patients with localized disease proceed to definitive treatment as determined by the treating physician starting 2-4 weeks after the first injection.

After completion of study treatment, patients are followed up at weeks 4-8 (for patients who received definitive treatment) or 12 (for patients with unresectable disease) and then annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy-confirmed Merkel cell carcinoma
* Patients must have at least one injectable lesion, defined as an easily palpable superficial lesion (cutaneous, subcutaneous or lymph nodal metastasis) that can be accurately localized, stabilized by palpation, and is superficial enough to enable intratumoral injection and electroporation; the injectable lesion must not be in close proximity to another tissue (e.g. nerve, bone) that could put patient safety at risk
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 to 2
* Life expectancy of greater than three months
* Absolute neutrophil count > 1,000/uL
* Platelet count > 50,000/uL
* Creatinine =< 2.0 x upper limit of normal (ULN)
* Bilirubin =< 2.0 x ULN
* Prothrombin time (PT) and partial thromboplastin time (PTT) =< 1.5 x ULN
* Patients must be willing, at the time of the entry to the study, to undergo the pre-treatment fine needle aspiration (FNA) plus biopsy (if indicated) AND the post-treatment FNA plus biopsy (or surgery) of at least one injected lesion (FNA is essential to determine the primary endpoint of the study); NOTE: The pre-treatment biopsy will be obtained from a superficial not-to-be-injected lesion; the post-treatment biopsy of an injected lesion will be obviated if definitive surgical resection is planned
* The effects of this treatment approach on the developing human fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients must have the ability to understand and the willingness to sign a written informed consent document
* Both men and women, and members of all races and ethnic groups are eligible for this trial

Exclusion Criteria:

* Patients who have had prior chemotherapy, investigational therapy or a major surgical procedure within 4 weeks or radiotherapy within 2 weeks prior to first day of treatment
* Patients must not be receiving concurrently any other anti-cancer treatment (including topical agents such as imiquimod) or investigational agents, which could potentially interfere with the study treatment and/or study endpoints
* Patients with active untreated brain metastases will be excluded
* Pregnant or breast feeding women are excluded because effects of this treatment on the fetus or passage through milk are unknown
* Patients with electronic pacemakers or defibrillators or those with a history of life threatening cardiac arrhythmia or uncontrolled seizure disorder are excluded
* Use of any immunosuppressive treatments including corticosteroids, cyclosporine, mycophenolate mofetil et cetera, within 4 weeks prior to Day 1 of treatment will not be allowed; NOTE: Patients on topical or physiologic doses (for hormone-replacement therapy) of corticosteroids will be allowed
* Patients, who are judged to be immunosuppressed due to uncontrolled human immunodeficiency virus (HIV) infection, severe uncontrolled diabetes, concurrent hematological malignancy, or other comorbidities, will be excluded
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active serious infection, symptomatic congestive heart failure, unstable angina pectoris, serious autoimmune conditions or psychiatric illness/social situations that would limit compliance with study requirements
* Patients receiving concurrent therapeutic-dose anticoagulation will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-01-03 (Actual); Primary Completion 2015-04-10 (Actual); Study Completion 2015-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shailender Bhatia, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 1 investigative site in the United States from 03 January 2012 to 10 April 2015.
Groups:
- Cohort B: Tavo-EP: Patients in Cohort B received up to 4 cycles (3 daily treatments on Days 1, 5, and 8, per cycle) of intra-tumoral injection(s) of tavo at a fixed dose of 0.5 mg/mL (up to 4 tumor sites) followed immediately by in vivo electroporation, with 12 weeks planned between each cycle, lasting up to 12 months.
Period: Overall Study
Arm/Group | Cohort A: Tavo-EP | Cohort B: Tavo-EP
Started | 3 | 12
Completed | 2 | 1
Not Completed | 1 | 11
Not completed — Disease Progression | 0 | 9
Not completed — To Be Seen By Local Oncologist | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, all patients who received any amount of the study drug (tavo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Tavo-EP | Cohort B: Tavo-EP | Total
Number analyzed (Participants) | 3 | 12 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (11.59) | 68.7 (12.08) | 67.1 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 3 | 9 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 12 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced At Least 2-Fold Increase in Expression of IL-12 Protein in the Tumor Tissue After Intratumoral (IT) pIL-12 Injections and In Vivo Electroporation
Description: The MAGPIX assay was used to assess differential expression of hIL-12 in patient tumor tissue before and after treatment with intratumoral (IT) tavo injections and in vivo electroporation (EP). Expression of hIL-12 was used to identify patients who met the primary endpoint of a 2-fold or higher increase in expression of hIL-12 in tumors after treatment. Fold change was taken as a comparison of hIL-12 expression at Week 3:pre-treatment, Week 6:pre-treatment, Week 8:pre-treatment, or Week 13:pre-treatment over baseline (pre- treatment). The fold change was calculated as log2 (time point/baseline).
Time Frame: Pre-treatment up to Week 13
Population: Efficacy Analysis Set, all patients from Cohort B who received any amount of the study drug (tavo).
Measure: Number; unit: percentage of participants
Arm/Group | Cohort B: Tavo-EP
Number analyzed (Participants) | 12
percentage of participants | 83

2. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, medical treatment or procedure and which did not necessarily have to have had a causal relationship with this treatment. An adverse event could have, therefore, been any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, medical treatment or procedure whether or not considered related to the medicinal product. An SAE was defined an any untoward medical occurrence that at any dosage resulted in one or more of the following: death, A life-threatening adverse event (real risk of dying), inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly, required intervention to prevent permanent impairment of damage.
Time Frame: From signing of informed consent to 8 weeks after the last dose of study treatment (up to 15 months)
Population: Safety Analysis Set, all patients who received any amount of the study drug (tavo).
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Tavo-EP | Cohort B: Tavo-EP
Number analyzed (Participants) | 3 | 12
percentage of participants
  AEs | 100 | 100
  SAEs | 0 | 8.3

3. Secondary Outcome: Objective Response Rate (ORR) in Injected and Non-injected (Distant) Lesions
Description: ORR is defined as the percentage of participants with evaluable lesions that achieved a complete response (CR) or partial response (PR) as assessed by the investigator using Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR: Disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: At least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions.
  The same method was used to assess response rate for treated lesions and response rate for non-treated lesions. The best response rate for non-treated lesions was based on the number of patients who had at least one non-treated lesion.
Time Frame: 3-4 weeks after the first dose in each cycle and then every 3 months until disease progression, death or withdrawal of consent (up to 15 months)
Population: Efficacy Analysis Set, all patients from Cohort B who received any amount of the study drug (tavo) and had evaluable lesions.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort B: Tavo-EP
Number analyzed (Participants) | 12
percentage of participants
  Injected Lesions: number analyzed (Participants) | 9
  Injected Lesions | 33.3
  Non-Injected Lesions: number analyzed (Participants) | 10
  Non-Injected Lesions | 20.0

4. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the number of days between the treatment initiation date (Study Day 1) and the earliest date of documented disease progression as defined by RECIST 1.1 or death that is not associated with prior disease progression. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: as for outcome 3
Population: Efficacy Analysis Set, all patients from Cohort B who received any amount of the study drug (tavo) and had document disease progression.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort B: Tavo-EP
Number analyzed (Participants) | 10
days | 52.5 [42.0 to 84.0]

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time in days from the date of first study drug administration to the date of death.
Time Frame: From the start of study treatment until death (up to 15 months)
Population: Efficacy Analysis Set, all patients who received any amount of the study drug (tavo). Zero participants were analyzed for overall survival because all patients were alive at their study completion visit.
Arm/Group | Cohort A: Tavo-EP | Cohort B: Tavo-EP
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Immunologic Effects of IT pIL-12 Injection and In Vivo EP Measured By: Percentage of Participants With a Positive Fold Change (Log2) in IL-12A Messenger Ribonucleic Acid (mRNA) for Patient Pre- and Post IT pIL 12 EP
Description: Nanostring analysis was performed to determine the expression (mRNA) of IL-12. For each study patient, the fold change (log2 transformed) in IL-12A mRNA as measured by Nanostring was determined using the pre-treatment (screening) biopsy as a reference for the post treatment biopsy. A log2 fold change >=1 is a positive result.
Time Frame: Pre-treatment up to Week 13
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort B: Tavo-EP
Number analyzed (Participants) | 6
percentage of participants | 66.6

7. Secondary Outcome: Local Regression Rate
Description: Local regression rate is defined as the percentage of participants with ≥30% regression (decrease in size) of at least one assessed local (injected) lesion.
Time Frame: as for outcome 3
Population: All patients from Cohorts A and B with evaluable lesions.
Measure: Number; unit: percentage of participants
Groups:
- All Patients: Tavo-EP: All patients from Cohort A and Cohort B.
Arm/Group | All Patients: Tavo-EP
Number analyzed (Participants) | 15
percentage of participants | 45.5

8. Secondary Outcome: Distant Regression Rate
Description: Distant regression rate is defined as the percentage of participants with ≥30% regression (decrease in size) of at least one assessed distant (non-injected) lesion.
Time Frame: as for outcome 3
Population: All patients from Cohorts A and B with evaluable lesions.
Measure: Number; unit: percentage of participants
Arm/Group | All Patients: Tavo-EP
Number analyzed (Participants) | 12
percentage of participants | 22.2

ADVERSE EVENTS:
Time Frame: From signing of informed consent to 8 weeks after the last dose of study treatment (up to 15 months).
Arm/Group | Cohort A: Tavo-EP | Cohort B: Tavo-EP
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/12
Other Adverse Events (participants affected / at risk) | 3/3 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Tavo-EP (N=3) | Cohort B: Tavo-EP (N=12)
Urinary tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Tavo-EP (N=3) | Cohort B: Tavo-EP (N=12)
Procedural pain (Injury, poisoning and procedural complications) | 3 | 12
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Injection site inflammation (General disorders) | 2 | 6
Injection site discolouration (General disorders) | 1 | 4
Fatigue (General disorders) | 0 | 3
Injection site bruising (General disorders) | 1 | 2
Injection site erythema (General disorders) | 0 | 1
Injection site haematoma (General disorders) | 1 | 0
Injection site necrosis (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Injection site cellulitis (Infections and infestations) | 1 | 2
Lung infection (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less